CLINICAL TRIAL: NCT06224361
Title: Reliability of a New Balance Assessment System in Patients With Adolescent Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elcin Akyurek, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: AkyurekE2
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Scoliosis; Adolescence
Keywords: scoliosis; postural control; balance; reliability
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Reliability: Participants will be evaluated with the "Postural Stability Test", "Limits of Stability Test", "Sensory Integration Test" and "Bilateral Comparison Test" within the AlBalance Balance Evaluation System. To calculate the test-retest reliability of the device, these measurements will be made by the same evaluator, will last 30 seconds and will be repeated a total of 3 times with a 1-minute rest between tests. These measurements will be repeated after 7 days to evaluate reliability. Then, parallel clinical tests will be applied to the participants, "Functional Reaching Test" and "One Leg Standing Test".

SUMMARY:
Postural stability is one of the most important factors that determine a person's ability to make and maintain movements. It has been reported that in the presence of scoliosis, the postural stability of people is negatively affected due to somatosensory disorders. There are many studies in the literature that evaluate the postural stability of cases diagnosed with scoliosis with objective methods. Evaluation of postural oscillations with objective devices is used to determine whether postural stability changes in AIS and whether the type and location of scoliosis affect the progression. The most commonly used objective devices for this purpose are balanced assessment systems in which changes in postural sway are recorded on the force platform. Our study aims to investigate the reliability of the "Postural Stability", "Limits of Stability", "Sensory Integration" and "Bilateral Comparison" tests of the Al Balance Balance Exercise and Analysis System in cases with Adolescent Idiopathic Scoliosis. After the demographic information of the cases that meet the inclusion criteria within the scope of the study is recorded, postural stability and balance evaluations within the Al Balance System will be performed on the cases. Evaluations will be carried out with bare feet and feet positioned at the same coordinates.

The tests will last 30 seconds and the test will be repeated a total of 3 times with a 1-minute rest between tests. These measurements will be repeated after 7 days to evaluate reliability.

With this study, the reliability of a new and local balance assessment system will be tested in cases with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12 and 18
* Having been diagnosed with Adolescent Idiopathic Scoliosis by an orthopedic specialist
* Cobb angle measured on anteroposterior radiograph is below 40 degrees
* Ability to understand and follow instructions
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of neuromuscular, rheumatic disease, or vestibular problems that may affect balance, vision-related diseases
* Having a recent history of orthopedic injury or surgery in the lower extremity
* Having had spine surgery
* Not having experienced any acute situation that could affect postural stability and balance between the two tests (within 7 days)
* Corset use has not changed between two tests (within 7 days)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents diagnosed with adolescent idiopathic scoliosis between the ages of 12-18 who meet the inclusion criteria will be included in our study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Postural Stability Test | Change from baseline to 7 day
  Stability indices represent fluctuations around the zero point established before testing when the platform is stable. With the "Postural Stability Test", the anteroposterior, right-left, and general stability indexes of the cases will be recorded. During the test, participants will be asked to stand on the force platform with their feet in a comfortable position, arms at their sides, and palms facing toward the thighs. All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. The participant will be asked to stand still looking at the screen in front of him for 30 seconds. There will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's Postural Stability will be assessed with Postural Stability Test.
Limits of Stability | Change from baseline to 7 day
  In this test, the participant stands on force plates and deliberately shifts his or her body weight in the direction indicated on the screen without lifting his or her feet off the ground. This protocol measures various movement characteristics in 8 different directions: front, forward/right, right, back/right, back, back/left, left, and forward/left. During the test, participants will be asked to stand on the force platform with their feet in a comfortable position, arms at their sides, and palms facing toward the thighs. Direction control (%) and test times (sec) in all directions of the participants, who will move in 8 different directions sequentially, will be recorded. There will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's Limits of Stability will be assessed with Limits of Stability Test.
Sensory Integration Test | Change from baseline to 7 day
  The test decides which of the visual, vestibular, and proprioceptive information is used to provide orientation to maintain balance in different situations. During the test, visual and proprioceptive stimuli are disrupted and the ability to maintain the center of gravity is evaluated. The test consists of 4 different situations that gradually become more difficult: Situation 1: Eyes open; firm surface Situation 2: Eyes closed; firm surface Situation 3: Eyes open; foam surface Situation 4: Eyes closed; foam surface All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. The participant will be asked to stand still looking at the screen in front of him for 30 seconds. There will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's Sensory Integration will be assessed with Sensory Integration Test.
Bilateral Comparison Test | Change from baseline to 7 day
  Bilateral Comparison test demonstrates postural stability by measuring the individual's ability to stand on one leg with eyes open and closed. On the balance platform, the individual stands on one leg with his hands at hip level. The test is repeated for the right foot and left foot. For both feet, 3 trials with eyes open and 3 trials with eyes closed are made. Each trial lasts 30 seconds. What is required from the individual is to remain stable on one leg as much as possible without losing balance. All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. The participant's Bilateral Comparison will be assessed with Bilateral Comparison Test.
Multimodal Functional Reach Test | Change from baseline to 7 day
  Multimodal functional reaching test is performed in three different positions: front, back, and side.
  In the functional forward reach test, the patient stands with the arm flexed at 90° and the fist closed, not touching but close to the wall. Three attempts are made and the average of these attempts is taken.
  In the functional back reach test, the patient stands with the arm flexed at 90° and the fist closed, not touching but close to the wall. Three attempts are made and the average of these attempts is taken.
  In the functional lateral reach test, the patient stands with his back to the wall, without touching the wall, keeping his arm in 90° abduction and his fist closed. Three attempts are made and the average of these attempts is taken. The participant's Multimodal Functional Reach balance will be assessed with Multimodal Functional Reach Test.
One Leg Stance Test | Change from baseline to 7 day
  The one-leg stance test demonstrates postural stability by measuring the individual's ability to stand on one leg with eyes open and closed. The individual stands on one leg with his hands at hip level. The test is repeated for the right foot and left foot. For both feet, 3 trials with eyes open and 3 trials with eyes closed are made. Each trial lasts 30 seconds. What is required from the individual is to remain stable on one leg as much as possible without losing balance. The participant's One Leg Stance balance will be assessed with One Leg Stance Test.

CONTACTS AND LOCATIONS:
Overall Officials: Asena Yekdaneh, Principal Investigator — Fenerbahçe University; İrem Kurt Ulusoy, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Nilay Arman, Principal Investigator — Istanbul University-Cerrahpasa Faculty of Health Science; Ayşe Zengin Alpözgen, Principal Investigator — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Elçin Akyürek, Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education